CLINICAL TRIAL: NCT02910336
Title: Somatosensory Investigation of Orofacial Pain Patients
Acronym: QST
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Galhardoni, PhD, University of Sao Paulo
Other Study IDs: MYTP-01
Record Dates: First submitted 2016-03-31; First posted 2016-09-22 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Facial Pain; Comorbidity; Neuralgia
MeSH Terms: conditions — Facial Pain; Neuralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Orofacial Pain patients under went to quantitative sensory test
  Interventions: Other: Quantitative Sensory Testing
- Control: Volunteers and presented neither previous diagnostic of orofacial pain nor generalized pain, under went to quantitative sensory test
  Interventions: Other: Quantitative Sensory Testing

INTERVENTIONS:
Other: Quantitative Sensory Testing — sensory testing profile

SUMMARY:
Orofacial pain, specially neuropathic orofacial pain, is a challenge of diagnosis and treatment in orofacial pain. It is associated with sensory abnormalities.With increasing life expectancy of the population is more and more common to find individuals with chronic diseases however, there is little evidence about the influence of comorbidities and medications in use on sensory thresholds of neuropathic orofacial pain. Objective: to investigate the influence of comorbidities and medication in somatosensory function of patients with orofacial neuropathic pain compared to controls.In this case-control study, 336 orofacial pain patients and controls were recruited from the Hospital das Clinicas da Faculdade de Medicina da USP were investigated about comorbidities, use of chronic medication, pain characteristics and a detailed standardized protocol of somatosensory evaluation at the trigeminal territories for cold, warm, tactile, vibration, deep, superficial and electric pain thresholds.

DETAILED DESCRIPTION:
Comorbidities The patients were interviewed by the same orofacial pain specialist using a questioner at the moment of the quantitative sensitive test.

Orofacial evaluation Instruments for orofacial evaluation. The questionnaires and exams were performed by one researcher only, a dentist, who ensured the clear understanding of the content by the participants before starting the protocol. All subjects underwent a standardized protocol for the evaluation of the orofacial region, including main complaint, pain characteristics [location, quality, duration, descriptors, intensity by the Visual Analog Scale (VAS), alleviation and aggravation factors], earache, headache, generalized body pain, sleep disturbances. Masticatory complaints related to parafunctional habits, laterality and the quality of mastication were also investigated. The intensity of masticatory discomfort was evaluated with the VAS. The intraoral examination included the evaluation of teeth, periodontal tissues, oral mucosa, tongue, lips, and facial skin, prostheses, occlusion and functional aspects, such as mandibular movements (mouth opening, protrusion, laterality) and temporomandibular joint (TMJ) exam (noises, spontaneous pain, or pain concomitant with movements). The muscular palpation of the head and neck was performed at the bilateral masseter, temporalis, digastrics, sternocleidomastoid, trapezius, splenius and suboccipitals. The periodontal exam was performed with adequate probes and the diagnoses made in accordance to the criteria of the American Academy of Periodontology. All participants underwent this detailed investigation for differential diagnosis with dental pain etiologies. Previous studies have shown that they can be associated with the main diagnosis of the patients.

Sensory investigation All subjects were interviewed about their perception of sensorial abnormalities such as numbness, dysesthesia, taste and smell complaints. The frequency of these abnormalities (absent, eventual, frequent, or constant) and the intensity (0-10 by VAS) were analyzed. This protocol is important for neuropathic and non-neuropathic pain diseases because somatic pain also presents sensitization and chronification.

QST. All subjects underwent a standardized protocol of QST which consists of 8 tests grouped as follows:

* gustative and olfactory thresholds;
* thermal detection thresholds for cold and warm sensations;
* mechanical detection thresholds for touch and vibration;
* mechanical pain sensitivity including superficial and deep pain thresholds. The somatosensory testing was performed at the 3 trigeminal branches (ophthalmic: fronte2 cm above the pupil, maxillary: cheek e 1 cm lateral to the nose wing, and mandibular: chin skin e 1 cm below the lip angle), at the hand dorsum (1 cm lateral to the thumb basis) and the anterior tibia skin (10 cm below the basis of patella). The evaluation was performed bilaterally in all subjects. All subjects were evaluated in the sitting position, with the head resting at a flat surface, and in a silent room with acoustic protection and the door closed. Only the participant and the researcher were in the room. All subjects were evaluated by the same researcher. The participants were oriented to keep the eyes closed during the exam, to be focused on the stimuli, and to their location (face and mouth) and characteristics. Only the researcher knew the order of the stimuli. Gustative thresholds: the following four substances, corresponding to the 4 tastes, were tested. For each test, one drop was applied at the tongue, starting with the low concentration, interleaved with one drop of distillate water, and the concentrations were tested until the subject had detected and identified the stimulus.

Sweet: glucose (0.01 M; 0.032 M; 0.1 M; 0.32 M; 1.0 M); Salty: sodium chloride (0.01 M; 0.032 M; 0.1 M; 0.32 M;1.0 M); Sour: citric acid (0.00032 M; 0.001 M; 0.0032 M;0.01 M; 0.032 M); Bitter: urea (0.1 M; 0.32 M; 1.0 M;3.2 M; 10.0 M). Olfactory thresholds: the subjects were evaluated with isopropanol solutions in polyethylene bottles interleaved with distillate water, starting with the lowconcentration until the subject had detected the stimulus;0.09%, 13.0%, 23.0%, 35.0%, 53.0%, 70.0%.

Thermal detection: thermal testing was performed using the MSA thermo test device (Somedic, Sweden). The baseline temperature was 32°C and the contact square area of the thermode was 9 x 9 mm. Cold detection threshold and warm detection threshold were assessed using ramped stimuli 1°C/s. The evaluation consisted in 5 measurements for each thermal threshold, and the means and standard deviations were considered for the analysis.

Mechanical detection threshold: touch perception was assessed using a set of standardized von Frey filaments with rounded tips of 0.5 mm diameter, applied with an electronic device (IITC, Woodland Hills, CA, USA). Three measurements in g/mm2 were performed and the means and SDs were considered for the analysis.

Vibration detection threshold: vibration testing was was performed using the electronic Vibrameter device(Somedic, Sweden) with a vibrator of 650 g of weight and a contact area of 1 cm2 perpendicularly applied for the thresholds detection, using ramped stimuli of 1 Hz/s. The method of calculation of vibration threshold consisted in the mean between the appearance and disappearance thresholds detected by the patient.

Pressure pain perception: deep pain thresholds were measured with the electronic pressure algometer (Somedic, Sweden) with a probe area of 1 cm2 which was pressed on the skin with a ramp rate of 50 kPa/s. Superficial pain perception: superficial pain thresholds were determined using disposable needles of 8x10x0.5 mm, applied with an electronic device (IITC, Woodland Hills, CA, USA). Three measurements in g/mm2 were performed and the means and SDs were considered for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Cases are participants with orofacial pain for more than six months prior to the evaluation

Exclusion Criteria:

* Case and controls were excluded if they had any history of trauma on face and/or skull surgery (except post traumatic neuropathic pain), generalized pain (except fibromyalgia), systemic diseases that cause neuropathy, neurodegenerative diseases, neuroendocrine diseases (except Diabetes Mellitus), rheumatologic diseases, and neuroinfectious diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The orofacial pain conditions include neuropathic pain, Temporomandibular Disorders (TMD), headache and fibromyalgia were diagnosed according to IASP (International Association for the Study of Pain) criteria. TMD were diagnosed following the American Academy of Orofacial Pain (AAOP). All orofacial pain were diagnoses by a trained orofacial pain specialist. Finally, patients with headache were diagnosed by a neurologist using the International Headache Classification (ICHD) criteria. Diabetes mellitus and diabetic neuropathy were diagnosed by an endocrinologist from our Hospital according to the World Health Organization (WHO) recommendations and fibromyalgia were diagnosed by a physiatrist using the American Academy of Rheumatology criteria. All controls were healthy and presented neither previous diagnostic of orofacial pain nor generalized pain.
Sampling Method: Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Sensory abnormalities measure through quantitative sensory testing | base line: 2 hours examination
  Quantitative sensory testing was used to measure alteration in sensory profiles. We used to measure differences in a cohort of patients with neuropathic orofacial pain, different stimuli, such as: cold and warm detection threshold, cold and heat pain threshold, mechanical detection threshold, pain mechanical threshold and vibration detection.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Siqueira, DDS, PhD, Principal Investigator — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No